CLINICAL TRIAL: NCT03103646
Title: Interventional, Open-label, One-sequence Crossover Study Evaluating the Effect of Multiple Doses of Itraconazole (Inhibitor of CYP3A4/5) on the Pharmacokinetics, Safety and Tolerability of Lu AF35700 in Healthy Young Men and Women
Brief Title: Study Evaluating the Effect of Multiple Doses of Itraconazole on the Drug Lu AF35700 in Healthy Young Men and Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17208A; 2016-003302-14 (EudraCT Number)
Record Dates: First submitted 2017-03-31; First posted 2017-04-06 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-10

CONDITIONS: Cytochrome P450 Interaction
MeSH Terms: interventions — Lu AF35700; Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lu AF35700 (Experimental): Day 1: Single dose of Lu AF35700. Extensive metabolisers (EMs): 10mg. Poor metabolisers (PMs): 5 mg
  Interventions: Drug: Lu AF35700
- Lu AF35700 AND itraconazole (Experimental): Days 29 to 31: once-daily dosage of 200 mg itraconazole. Day 32: Single dose of Lu AF35700 (EMs: 10 mg, PMs: 5 mg) and 300 mg itraconazole Days 33 to 42: once-daily dosage of 200 mg itraconazole
  Interventions: Drug: Lu AF35700; Drug: Itraconazole (200 mg); Drug: Itraconazole (300 mg)

INTERVENTIONS:
Drug: Lu AF35700 — Tablets for oral use, single dose in a fasted state. EMs: 10 mg/day, PMs: 5 mg
Drug: Itraconazole (200 mg) — 100 mg Capsules for oral use, 200 mg/day. In a fed state
  Arms: Lu AF35700 AND itraconazole
Drug: Itraconazole (300 mg) — 100mg Capsules for oral use, 300 mg/day. In a fasted state.
  Arms: Lu AF35700 AND itraconazole

SUMMARY:
This study will investigate the effect of multiple doses of the strong P450 enzyme inhibitor itraconazole on the pharmacokinetics of Lu AF35700 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Men, aged ≥18 and ≤55 years. body weight ≥50 kg
* women, aged ≥18 and ≤45 years, body weight ≥50 kg
* Good general health as assessed using detailed medical history, laboratory tests, and physical examination
* Known CYP2D6 and CYP2C19 genotype

Exclusion Criteria:

* Pregnant or lactating
* Subject has previously been dosed with Lu AF35700

Other protocol defined inclusion and exclusion criteria may apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2017-03-28 (Actual); Primary Completion 2019-04-14 (Actual); Study Completion 2019-07-19 (Actual)

PRIMARY OUTCOMES:
AUC(0-inf) | Day 1: Predose to day 29 postdose, Day 32: Predose to day 74 postdose
  Area under the Lu AF35700 plasma concentration-time curve (with and without itraconazole) for CYP2D6 EMs
Cmax | 0-24 hours postdose (Day 1 and day 32)
  Maximum observed plasma concentration of Lu AF35700 (with and without itraconazole) for CYP2D6 EMs

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@Lundbeck.com
Locations (2):
- Covance - Dallas, Dallas, Texas, United States
- Covance Clinical Research Unit Ltd, Leeds, United Kingdom